CLINICAL TRIAL: NCT02930382
Title: Assessment of Spontaneous Baroreflex Sensitivity in Carriers of Implantable Cardioverter Defibrillators: Association With Disorders of the Ventricular Heart Rate. Case-control Study
Acronym: BARODEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BARODEF
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

ARMS (1):
- BAROREFLEX (Experimental)
  Interventions: Other: Baroreflex assessment

INTERVENTIONS:
Other: Baroreflex assessment

SUMMARY:
We must implement 8 implantable cardioverter defibrillators (ICDs) to save a life in 3 years after myocardial infarction (MI) in primary prevention.

Left ventricular ejection fraction (LVEF) is proposed as the one tool predicting sudden cardiac death after MI.

Several studies have shown that impairment of spontaneous baroreflex sensitivity (BRS) after MI was predictor of sudden death.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with an implantable cardioverter defibrillator for primary prevention of of cardiac sudden death, ischaemic cardiomyopathy
* Implantable cardioverter defibrillators implantation for at least 3 years
* Age ≥ 18 years

Exclusion Criteria:

* ventricular or atrial pacing ≥1%,
* atrial fibrillation history
* age under 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

PRIMARY OUTCOMES:
spontaneous baroreflex sensitivity by the sequence method (mean slope) | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU DE Poitiers, Poitiers, France